CLINICAL TRIAL: NCT04064996
Title: Effectiveness of Foot Exercise Training on Patients With Type 2 Diabetes and Peripheral Neuropathy
Brief Title: Effectiveness of Foot Exercise People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Evrim KOÇARSLAN, physiotherapist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 199292
Record Dates: First submitted 2019-08-17; First posted 2019-08-22 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 2; Peripheral Neuropathy
Keywords: foot exercise; pain
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Nervous System Diseases; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Routine rehabilitation program patient education
  Interventions: Other: Routine rehabilitation program patient education
- Group B (Experimental): Routine rehabilitation program + foot exercise training
  Interventions: Other: Routine rehabilitation program + foot exercise training

INTERVENTIONS:
Other: Routine rehabilitation program patient education — Patient education
  All the patients were assessed with Wagner Classification, Diabetic Neuropathy Symptom (DNS) score, Diabetic Neuropathy Examination (DNE) score, Visual Analogue Scale (VAS), Leeds assessment of neuropathic symptoms and signs (LANSS), hand-held dynamometer, range of motion measurements, Semmes-Weinstein monofilament, two point discrimination test, circumference measurements, Foot and Ankle Ability Measure(FAAM), 6-minute walk test (6MWT) before and after the treatment.
  Arms: Group A
Other: Routine rehabilitation program + foot exercise training — In addition to the patient education , foot exercise training will be performed. Patients will be applied exercise training consisted of aerobic, strengthening, sensory training and stretching exercises for 3 days/week, 8 weeks.
  All the patients were assessed with Wagner Classification, Diabetic Neuropathy Symptom (DNS) score, Diabetic Neuropathy Examination (DNE) score, Visual Analogue Scale (VAS), Leeds assessment of neuropathic symptoms and signs (LANSS) ,hand-held dynamometer,range of motion measurements, Semmes-Weinstein monofilament, two point discrimination test,circumference measurements, Foot and Ankle Ability Measure(FAAM), 6-minute walk test (6MWT) before and after the treatment.
  Arms: Group B

SUMMARY:
The aim of this study will to investigate the effect of foot exercises in patients with type 2 diabetic and peripheral neuropathy. Subjects will be randomly allocated to either the control or intervention group. Data will be collected using investigator-developed forms: patient information form and the diabetic foot exercises log. Patients in the intervention group will be received standard treatment and performed foot exercises for three times a week 8 weeks; the control group will be received standard treatment but no exercises. The intervention and control groups will be examined and measured at the 4th and 8th weeks.

DETAILED DESCRIPTION:
Purpose of our study investigation of the effects foot exercises in patients with type 2 diabetic and peripheral neuropathy.

Excepted results: Routine treatment + foot exercises pain, flexibility, edema, muscle strength, sensation, quality of life we believe that there will be good progress in peripheral neuropathy effects, Leeds assessment of neuropathic symptoms and signs(LANSS) results.

In this context, it is planned that patients randomly divided into 2 groups. Group 1 control group. Group 2 intervention group. Patients in the intervention group will be received standard treatment and performed foot exercises for three times a week 8 weeks. The patients will be evaluated by clinical measurements and scales based on patient notification at the 4th and 8th weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having type 2 diabetes mellitus for 5 years
* HbA1c > among of between 6.5-10
* Having grade 0 or 1 phase of Wagner classification
* Diabetic neuropathy score ≥ 3

Exclusion Criteria:

* Not to know turkish
* Having hearing, visual and speaking problems
* Having (except diabetic neuropathy) other neurologic problems
* Having psychiatric and cognitive problems
* Having orthopedic, rheumatologic, cardiac, and pulmonary problems which stopping exercise

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Pain assessment with Algometry | Change from Baseline Pain at 8 weeks
  An instrument for determining sensitivity to pain produced by pressure.
Pain assessment with The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale | Change from Baseline Pain at 8 weeks
  The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale evaluates sensory dysfunction and whether the pain is caused by neuropathic mechanisms or not. The LANSS comprises a 5-item questionnaire regarding pain symptoms and two items for clinical signs involving self-administered sensory tests for the presence of allodynia and decreased sensation to pinprick. Responses to each item are binary (yes or no) and each item is weighted differently depending on the odds ratio of a positive response to each item to predict that the pain is primarily neuropathic. The possible scores range from 0 to 24, with a score of 12 or greater considered to be suggestive of neuropathic pain
Pain assessment With Visual Analog Scale | Change from Baseline Pain at 8 weeks
  Participants are asked to mark the point where they feel their pain on a 10 centimeter (cm) horizontal line. 0-no pain, 10-unbearable pain. Night, activity and pain conditions are evaluated separately at rest.

SECONDARY OUTCOMES:
Muscle Strength with Hand held dynamometer | 1th day, 8th week
  The Hand-Held Dynamometer (formerly known as the Manual Muscle Tester) is an ergonomic hand-held device for objectively quantifying muscle strength.
Range Of Motion with goniometer | 1th day, 8th week
  A goniometer is a device used in physical therapy to measure the range of motion around a joint in the body.
Baseline Tactile Semmes-Weinstein Monofilament | 1th day, 8th week
  Baseline Tactile Semmes-Weinstein Monofilaments are designed to measure cutaneous sensory perception threshold of a patient.
Edema measurement of tape | 1th day, 8th week
  Use a measuring tape to measure the circumference of your leg. Write down its circumference and repeat daily for a few days, using the same area on your the leg.
Evaluation of functional capacity with 6 minutes walking test | 1th day, 8th week
  The 6-minute walk test is one of the functional exercise capacity assessment tests. In this test, participants are asked to walk as long as possible within 6 minutes in a 30 meter (m) corridor. When they feel fatigue or pain, they are advised to stop and rest when they feel ready to walk. At the end of 6 minutes, the total distance of the patients walking is recorded. Heart rates, systolic and diastolic blood pressures, O2 saturation, perceived fatigue and dyspnea levels are recorded before and after the test.
Two Point Discrimation Test | 1th day, 8th week
  The two-point discrimination test is used to assess if the patient is able to identify two close points on a small area of skin, and how fine the ability to discriminate this are. It is a measure of tactile agnosia, or the inability to recognize these two points despite intact cutaneous sensation and proprioception.
The Foot and Ankle Ability Measure | 1th day, 8th week
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments.
HbA1c | 1 th day, 8th week
  HbA1c (A1c or glycosylated hemoglobin) is widely used as the most important marker for routine monitoring of long term glycemic status in patients with diabetes.
Serum creatinine | 1 th day, 8th week
  The kidneys are responsible for keeping the level of creatinine in the blood within a normal range. The typical reference range for serum creatinine is 60 to 110 micromoles per liter (μmol/L) (0.7 to 1.2 milligrams per deciliter (mg/dL)) for men and 45 to 90 μmol/L (0.5 to 1.0 mg/dL) for women.
Albumin levels | 1 th day, 8th week
  A normal albumin range is 3.4 to 5.4 g/dL. If you have a lower albumin level, you may have malnutrition. It can also mean that you have liver disease or an inflammatory disease. Higher albumin levels may be caused by acute infections, burns, and stress from surgery or a heart attack.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Koçarslan, Principal Investigator — researcher
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Francia P, Gulisano M, Anichini R, Seghieri G. Diabetic foot and exercise therapy: step by step the role of rigid posture and biomechanics treatment. Curr Diabetes Rev. 2014 Mar;10(2):86-99. doi: 10.2174/1573399810666140507112536. PMID 24807636